CLINICAL TRIAL: NCT03939299
Title: Optical Coherence Tomography Imaging Explores Long-term vasculAR Response and Healing profIle After successFul coronarY Stenting in Chronic Total Occlusion
Brief Title: OCT Explores Vascular Response and Healing Profile After Stenting in CTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLARIFY-CTO
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: subintimal stenting; vascular response and healing; optical coherence tomography

STUDY DESIGN:
Intervention Model Description: All enrolled patients received optical coherence tomography examination after successful stening at the chronic total occlusion lesion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCT group (Experimental): Patients, whose coronary chronic total occlusion lesion was successfully implanted stent, received optical coherence tomography imaging immediately and at 9-12 months after index procedure.
  Interventions: Procedure: OCT

INTERVENTIONS:
Procedure: OCT — Patients with coronary chronic total occlusion received successful stenting. Optimal coherence tomography imaged immediately and at 9-12 months after the index procedure to explore long-term vascular response and healing profile.

SUMMARY:
True-false-true occurred during wire penetration in coronary CTO procedure. Subintimal stenting influences vascular response. Intravenous ultrasound confirmed wire position in the procedure. Then stenting procedure was performed. Optical coherence tomography was used for exploring long-term vascular response and healing profile after successful coronary stenting in CTO lesions.

DETAILED DESCRIPTION:
Chronic total occlusions (CTOs) are defined as coronary lesions with thrombolysis in myocardial infarction (TIMI) grade flow of 0 and present for more than 3 months. CTO is commonly recognized as the toughest lesion subset to be treated by percutaneous coronary interventions. With the remarkable progress in the technologies and techniques achieved in the PCI for CTO over the last decade, the rate of procedural success increased to 80-90%. Chronic total occlusion is associated with a higher incidence of malapposition and uncovered stent struts. At present, four strategies were used for CTO lesions, including: ante-grade wire escalation, ante-grade dissection reentry (ADR), retro-grade wire escalation, and retrograde dissection reentry (RDR). True-false-true occurred during wire penetration. Subintimal stenting influences vascular response. Intravenous ultrasound (IVUS) confirmed wire position in the procedure. Then stenting procedure was performed according to standard routine. Optical coherence tomography (OCT) was used for exploring long-term vascular response and healing profile after successful coronary stenting in CTO lesions.

ELIGIBILITY:
Inclusion Criteria:

* 18~85 years old;
* Agree percutaneous coronary intervention without related contraindications;
* Chronic total occlusion confirmed by clinical and angiographic data, predicted high successful rate of stent implantation;
* Subjects (or legal guardians) understanding the testing requirements and procedures, and providing written informed consent.

Exclusion Criteria:

* Subjects associated with drugs allergy (such as contrast, sirolimus, or structure-related compounds fluorinated polymers, thienopyridine or aspirin);
* Subjects with active peptic ulcer, active gastrointestinal (GI) bleeding or other bleeding diathesis or coagulopathy;
* Subjects being suffered from other serious illness (such as cancer, congestive heart failure), which may cause drop in life expectancy to less than 12 months;
* Pregnant or breastfeeding women;
* Refused this trial;
* Subjects with severe liver or renal dysfunction (ALT >5×ULN，eGFR< 30ml/min/1.73mm2 or Scr>200 mmol/L);
* Active bleeding;
* Bleeding diathesis or coagulopathy, malignant tumors;
* Contraindication of anticoagulant drugs;
* Subjects with other situation not suitable for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
long-term minimal stent area | 9-12 month after index procedure
  measured through OCT imaging result
long-term stent thrombosis | 9-12 month after index procedure
  measured through OCT imaging result
long-term stent neointima | 9-12 month after index procedure
  measured through OCT imaging result
long-term stent malapposition | 9-12 month after index procedure
  measured through OCT imaging result
immediately minimal stent area | in the procedure
  measured through OCT imaging result
immediately stent malapposition | in the procedure
  measured through OCT imaging result

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events | 9-12 month after index procedure
  clinical follow-up record

CONTACTS AND LOCATIONS:
Overall Officials: Juying Qian, Professor, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China